CLINICAL TRIAL: NCT06619899
Title: Investigation of Post-activation Potentiation Phenomenon οn Sprinting Performance Following Power Pre-conditioning Exercise
Brief Title: Post-activation Potentiation and Sprinting Performance
Acronym: PAP-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: PAP-Sprinting
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sprint Performance
Keywords: post-activation potentiation; sprinting performance; power pre-conditioning exercise; speed
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PAP exercise with 0% body mass (Experimental): The participants will perform 6 x 30m sprints. A pre-conditioning exercise (2 sets x 4 countermovement jumps with 0% body mass).
  Interventions: Other: PAP exercise with 0% body mass
- PAP exercise with 20% body mass (Experimental): The participants will perform 6 x 30m sprints. A pre-conditioning exercise (2 sets x 4 countermovement jumps with 20% body mass).
  Interventions: Other: PAP exercise with 20% body mass
- No PAP exercise (Placebo Comparator): The participants will perform only 6 x 30m sprints. No pre-conditioning exercise will be performed.
  Interventions: Other: No PAP exercise

INTERVENTIONS:
Other: PAP exercise with 0% body mass — The participants will perform 6 x 30m sprints. Before each sprint they will perform 2 x 4 countermovement jumps with 0% body mass.
  Other Names: post-activation potentiation training; sprint training
  Arms: PAP exercise with 0% body mass
Other: PAP exercise with 20% body mass — Description: The participants will perform 6 x 30m sprints. Before each sprint they will perform 2 x 4 countermovement jumps with 0% body mass
  Other Names: post-activation potentiation training; sprint training
  Arms: PAP exercise with 20% body mass
Other: No PAP exercise — No PAP exercise will be performed. The participants will perform only 6 x 30m sprints.
  Other Names: post-activation potentiation training; sprint training
  Arms: No PAP exercise

SUMMARY:
Scientific data regarding the post-activation potentiation (PAP) phenomenon on sprinting performance is scarce, especially regarding the effect of performing pre-conditioning power exercises on subsequent sprinting performance. Additionally, there is no data regarding the rate of fatigue onset when power pre-conditioning exercise before sprints are performed repeatedly at the same training session. This research will provide important information to coaches and athletes for the design of an optimum training program for the maximization of the athletes' performance and the avoidance of injuries.

DETAILED DESCRIPTION:
Sprinting ability is an imperative quality for many sports, especially for sprint and power athletes. Regular sprint training improves acceleration, maximal speed and power. Thus, sprint training consists one of the basic elements of the athletes' training program.

One method used by coaches to improve performance is the implementation of a pre-conditioning exercise aiming to post-activation potentiation (PAP). Post-activation potentiation phenomenon refers to the increase in performance following a maximal or near maximal muscle contraction (e.g. a pre-conditioning exercise). However, the effectiveness of such an approach is under debate, such that improvement, but also no improvement, or even deterioration of the performance following pre-conditioning exercises has been reported. The improvement of performance following a pre-conditioning exercise seems to depend on the relationship between muscle twitch potentiation and fatigue following the pre-conditioning exercise. When muscle twitch potentiation is greater than muscle fatigue, then the PAP mechanism will be activated and performance will be improved. Contrary, under similar muscle twitch potentiation and fatigue, performance will not change, and when muscle twitch potentiation is lower than fatigue, muscle performance will decrease. PAP phenomenon has been studied mainly regarding its effectiveness to improve jumping performance, while its effectiveness on improving sprinting performance has not been adequately studied. However, information regarding the effectiveness of the implementation of pre-conditioning exercises aiming to improve sprinting performance, is important for the design of an optimum training program for the maximization of the athletes' performance and the avoidance of injuries.

The aim of this study is to investigate a) the effectiveness of the implementation of a pre-conditioning exercise to activate the PAP mechanism and improve performance of a following sprint, and b) to investigate whether PAP is maintained in repeated efforts during the same training session.

The study will be implemented in a randomized, cross over, repeated measures design, at three cycles.

According to a preliminary power analysis (a probability error of 0.05, and a statistical power of 80%), a sample size of 8 - 10 participants was considered appropriate in order to detect statistically meaningful differences between groups. Considering a possible drop-out, 15 participants will be recruited. Procedures will be in accordance with the 1964 Declaration of Helsinki, as revised in 2013.

Before the experimental procedures, all participants will sign an informed consent form after they will be informed about all the benefits and risks of the study, and they will also fill in a medical history questionnaire. Participants will then perform baseline measurements at the Laboratory of Biochemistry, Physiology and Nutrition of Exercise (SmArT Lab), Department of Physical Education and Sport Science, University of Thessaly: anthropometric characteristics (body height, body mass, body mass index) via a stadiometer-scale (Stadiometer 208; Seca, Birmingham, UK), body composition (percent of body fat, lean body mass, fat mass, bone density) via dual emission X-ray absorptiometry (DXA, GE-Healthcare, Lunar DPX NT, Belgium), isokinetic strength (isometric, concentric and eccentric torque of the knee extensors and knee flexors of both limbs) on an isokinetic dynamometer (Cybex, HUMAC NORM 360, Ronkonkoma, NY). The individual optimum rest period between the pre-conditioning exercise and the subsequent 30-m sprint will be estimated, in order each participant to perfrom each 30-m sprint under an optimal condition. The rest periods of 3, 6, and 9 minutes will be tested for each participant and the rest period that leads to the best sprinting performance will be applied during the experimental training protocols.

Participants will then perform 6 x 30-m sprints under three different conditions in a random order: a) control trial (sprint training without pre-conditioning exercise), b) sprint training with pre-conditioning exercise (2 x 4 squat jumps with 0% of 1RM at squat), and c) sprint training with pre-conditioning exercise (2 x 4 squat jumps with 20% of 1RM at squat). The randomization of the trials will be made via a random integer set generator (Random.org) available online.

Prior to, and following each 30-m sprint, assessment of muscle soreness in the knee flexors and knee extensors, countermovement jump height, and blood lactate concentration, will be performed during each training session. The exact above procedures will be repeated by the participants during the remaining two experimental trials. Between trials, a wash-out period of 7 days will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 30 years old
* Srinters or athletes that comprise sprint training in their training programs
* Absense of musculoskeletal injuries (≥ 6 months)
* Abstence from use of ergogenic supplements or other drugs (≥ 1 month)
* Abstence from participation at exercise with eccentric component (≥ 3 days)
* Abstence from alcohol and energy drings consumption before each experimental trial

Exclusion Criteria:

* Age: Older than 18 - 30 years
* Musculoskeletal injuries (≤ 6 months)
* Use of ergogenic supplements or other drugs (≤ 1 month)
* Participation at exercise with eccentric component (≤ 3 days)
* Alcohol and energy drings consumption before the experimental trials

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in 30 m sprint performance | Pre, 9, 18, 27, 36, and 45 minutes during the sprint training session.
  30-m sprint performance will be assessed via photocells.

SECONDARY OUTCOMES:
Changes in muscle soreness in the knee flexors and extensors of both limbs | Pre, 9, 18, 27, 36, and 45 minutes during the sprint training session.
  Muscle soreness will be assessed immediately post each 30-m sprint. Muscle soreness will be assessed via palpation of the muscle belly and the distal regions following 3 squats, and the subjective pain will be recorded on a 10-point scale (1 = no pain, 10 = extreme pain)
Changes in countermovement jump performance | Pre, 12, 21, 30, 39, and 58 minutes during the sprint training session.
  Countermovement jump performance will be assessed 3 minutes post each 30-m sprint via an optical measurement system
Changes in lactate | Pre, 13, 22, 31, 40, and 49 minutes during the sprint training session.
  Lactate will be measured 4 minutes following each 30-m sprint via a lactate portable analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, Associate Professor, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz LB, Haff GG. Factors Modulating Post-Activation Potentiation of Jump, Sprint, Throw, and Upper-Body Ballistic Performances: A Systematic Review with Meta-Analysis. Sports Med. 2016 Feb;46(2):231-40. doi: 10.1007/s40279-015-0415-7. PMID 26508319
- [Background] Rassier DE, Macintosh BR. Coexistence of potentiation and fatigue in skeletal muscle. Braz J Med Biol Res. 2000 May;33(5):499-508. doi: 10.1590/s0100-879x2000000500003. PMID 10775880
- [Background] Hodgson M, Docherty D, Robbins D. Post-activation potentiation: underlying physiology and implications for motor performance. Sports Med. 2005;35(7):585-95. doi: 10.2165/00007256-200535070-00004. PMID 16026172
- [Background] Bridgett LA, Linthorne NP. Changes in long jump take-off technique with increasing run-up speed. J Sports Sci. 2006 Aug;24(8):889-97. doi: 10.1080/02640410500298040. PMID 16815784